CLINICAL TRIAL: NCT02035618
Title: Exercises Associated or Not With Manual Therapy Shoulder Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Paula Rezende Camargo, PT, PhD, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFSCar/CEP 270/2010
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercises and manual therapy (Experimental)
  Interventions: Other: Exercises; Other: Exercises + Manual Therapy
- Exercises (Active Comparator)
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Strengthening and stretching
Other: Exercises + Manual Therapy — Mobilization; massage; post-isometric relaxation; strengthening; stretching
  Arms: Exercises and manual therapy

SUMMARY:
Manual therapy combined with a protocol of therapeutic exercises will increase the beneficial effects on scapular kinematics, myofascial pain and function in subjects with shoulder impingement when compared to exercises only.

ELIGIBILITY:
Inclusion Criteria:

* history of non-traumatic onset of shoulder pain;
* painful arc during active elevation of the arm;
* one or more positive shoulder impingement tests (Neer, Hawkins and Jobe), or pain during passive or resisted external rotation of the arm at 90° of abduction;
* pain with palpation of the rotator cuff tendons;
* all subjects need also to be able to reach 150° of arm elevation as evaluated by visual observation.

Exclusion Criteria:

* limitation of glenohumeral internal and external rotation as indicative of adhesive capsulitis;
* body mass index > 28kg/m2 as the amount of subcutaneous tissue can compromise the quality of the signal increasing soft tissue artifact;
* numbness or tingling of the upper limb reproduced by cervical compression test;
* history of clavicle, scapula or humerus fracture;
* history of rotator cuff surgery;
* systemic illnesses;
* positive sulcus or apprehension tests as indicative of instability;
* positive drop arm test as indicative of full thickness tear;
* corticosteroid injection within 3 months prior to intervention, or physiotherapy within 6 months prior to intervention;
* depressive symptoms as evaluated by the Beck Depression Inventory score ( > 9 points) due to its influence on myofascial pain;
* allergy to tape.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Scapular kinematics | up to 3 months from the initial interview

REFERENCES:
- [Derived] Camargo PR, Alburquerque-Sendin F, Avila MA, Haik MN, Vieira A, Salvini TF. Effects of Stretching and Strengthening Exercises, With and Without Manual Therapy, on Scapular Kinematics, Function, and Pain in Individuals With Shoulder Impingement: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2015 Dec;45(12):984-97. doi: 10.2519/jospt.2015.5939. Epub 2015 Oct 15. PMID 26471852